CLINICAL TRIAL: NCT03346408
Title: Dependence on Analgesics in Chronic Non-cancer Pain: Comparison of the Perceptions of the Algologist Physician and the Perception of the Patient.
Brief Title: Dependence on Analgesics in Chronic Non-cancer Pain
Acronym: DISCORDANCE
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/17/0094; 2017-A01826-47 (Other: IDRCB)
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Pain, Chronic
Keywords: Analgesics
MeSH Terms: conditions — Chronic Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: data collection obtained from patient (self-questionnaire) and algologist physician (questionnaire).
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — patient (self-questionnaire) and algologist physician (questionnaire)

SUMMARY:
The identification of an addiction to opioid analgesics has become strong recommendation for the purpose of improving the clinical management of the patients. However, the success of the patient's clinical management, in terms of analgesia and treatment of drug dependence, rests on the acceptance of this management by the patient himself. The main objective of this study is to evaluate the factors associated to the discrepancy between the assessment of dependence on analgesic drugs by the algologist and the perception that the patient with non-cancer chronic pain has of this dependence.

DETAILED DESCRIPTION:
The long-term use of opioid analgesics for the treatment of chronic non-cancer pain exposes patients to the risk of developing drug dependence on these psychoactive drugs with loss of control of their use. In general medicine as well as in algology consultation, the identification of an addiction to opioid analgesics (and even misuse as a gateway to addiction) have thus become strong recommendations for the purpose of improving the management of the patients. However, the success of the patient's clinical management, in terms of analgesia and treatment of drug dependence, rests on the acceptance of this management by the patient himself.

The discrepancy between the assessment of drug dependence on analgesic drugs by the algologist and the perception that the patient has of this dependence will be investigated through a multicentre cross-sectional descriptive survey performed in pain treatment centres in France.

In addition to opioid analgesics, other pharmacological classes used for analgesic use will be investigated as they are concerned with the development of drug dependence. This is particularly the case for gabapentins.

ELIGIBILITY:
Inclusion Criteria:

* suffering from chronic non-cancer pain,
* taking at least one analgesic medication

Exclusion Criteria:

* Patient minor or major protected by the law (under tutelage),
* Patient with chronic pain of cancerous origin,
* Opposition of the patient to be included in the study,
* Patient not having the overall skills to complete a self-questionnaire: major difficulties in understanding the French language and / or reading / writing difficulties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physician and patients recruited in pain consultations and treatment structures
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2017-11-04 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
discrepancy between the assessment of dependence on analgesic drugs by the algologist and the perception of the patient | Baseline
  The patients will complete a self-questionnaire and the algologist physician will fill another questionnaire.

SECONDARY OUTCOMES:
Consumption drugs | Baseline
  Patient questionnaire for associated drug
Anxiety | Baseline
  Hospital Anxiety and Depression Scale (HAD Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Anne ROUSSIN, PharmD PhD, Principal Investigator — University Hospital, Toulouse
Locations (7):
- France (7):
  - University Hospital Bordeaux, Bordeaux
  - University Hospital Clermont-Ferrand, Clermont-Ferrand
  - University Hospital Limoges, Limoges
  - University Hospital Marseille, Marseille
  - University Hospital Montpellier, Montpellier
  - University Hospital Nice, Nice
  - University HospitalToulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roussin A, Cisse Z, Rousseau V, Roche G, Lestrade C, Cauchie A, Delage N, Donnet A, Van Obberghen E, Wood C, Lapeyre-Mestre M, Cantagrel N. Discordance between pain specialists and patients on the perception of dependence on pain medication: A multi-centre cross-sectional study. Therapie. 2024 Sep-Oct;79(5):543-551. doi: 10.1016/j.therap.2024.01.008. Epub 2024 Apr 12. PMID 38653623